CLINICAL TRIAL: NCT02427750
Title: A Phase II, Open-Label, Single-Arm, Multicenter Study to Evaluate the Safety and Immunogenicity of a Surface Antigen, Inactivated, Egg-Derived, Trivalent Influenza (Agrippal®) Virus Vaccine, Southern Hemisphere Formulation 2015, in Healthy Adults.
Brief Title: A Study to Evaluate Safety and Immunogenicity of Trivalent Influenza Vaccine, Formulation 2015 Southern Hemisphere, When Administered to Healthy Adult Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V71_40S
Record Dates: First submitted 2015-04-13; First posted 2015-04-28 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Human Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trivalent Influenza Vaccine (Experimental): One injection of Agrippal®
  Interventions: Biological: Aggripal®

INTERVENTIONS:
Biological: Aggripal® — TIV

SUMMARY:
The present study is designed to evaluate the safety and immunogenicity of trivalent, surface antigen, inactivated influenza vaccine in 2 age cohorts: 18 to ≤60 years and ≥61 years.

For the immunogenicity endpoint the antibody response to each influenza vaccine antigen will be evaluated by means of Single Radial Hemolysis (SRH) or Hemagglutination Inhibition (HI) at approximately 21 days post vaccination.

The vaccine composition will be based on the WHO recommended influenza strains for the 2015 Southern Hemisphere vaccine, and the data from this study are intended to support the use of this vaccine in future influenza seasons if the recommended vaccine composition remains the same.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals of 18 years of age and above on the day of informed consent.
2. Individuals who have voluntarily given written informed consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
3. Individuals who can comply with study procedures including follow-up.
4. Males or females of non-child bearing potential or females of childbearing potential who are using an effective birth control method which they intend to use for at least 30 days after the last study vaccination.

Exclusion Criteria:

1. Progressive, unstable or uncontrolled clinical conditions.
2. Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study.
3. Clinical conditions representing a contraindication to intramuscular vaccination and blood drawn.
4. Abnormal function of the immune system resulting from:

   * Clinical conditions,
   * Systemic administration of corticosteroids (PO/IV/IM) for more than 14 consecutive days within 90 days prior to informed consent,
   * Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent,
5. Received immunoglobulins or any blood products within 180 days prior to enrollment.
6. Received an investigational or non-registered medicinal product within 30 days prior to enrollment.
7. Study personnel as an immediate family or household member.
8. Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrolment in this study or who are planning to receive any vaccine within 28 days from the study vaccines.
9. Has behavioral or cognitive impairment, psychiatric disease, severe neurological (especially Guillain-Barré syndrome) that, in the opinion of the investigator may interfere with the subject's ability to participate in the study.
10. Has a serious chronic or acute disease (in the judgment of the investigator may interfere with the result of the study or pose additional risk to the subject) including but not limited to:

    * medically significant cancer (except for benign or localized skin cancer, cancer in remission for ≥10 years, or localized prostate cancer that has been clinically stable for >2 years without treatment),
    * medically significant advanced congestive heart failure (i.e., New York Heart Association [NYHA] class III and IV),
    * chronic obstructive pulmonary disease (ie, Global initiative for chronic Obstructive Lung Disease stage III and IV),
    * autoimmune disease (including rheumatoid arthritis and excepting Hashimoto's thyroiditis that has been clinically stable for ≥5 years),
    * diabetes mellitus type I,
    * poorly controlled diabetes mellitus type II,
    * advanced arteriosclerotic disease,
    * history of underlying medical condition such as major congenital abnormalities requiring surgery, chronic treatment, or associated with developmental delay (e.g., Down's syndrome),
    * acute or progressive hepatic disease,
    * acute or progressive renal disease,
    * severe asthma.
11. Has known or suspected drug or alcohol abuse within the past 2 years;
12. Has the following within the past 6 months:

    * had any laboratory-confirmed seasonal or pandemic influenza disease,
    * received any seasonal or pandemic influenza vaccine,
13. Has acute or chronic infections requiring systemic antibiotic treatment or antiviral therapy within the last 7 days;
14. Has experienced fever (i.e., body temperature [preferably axillary] ≥38.0°C) within the last 3 days of intended study vaccination;
15. Has a body mass index (BMI) >35 kg/m2 (BMI is calculated by dividing the subject's weight in kilograms by the subject's height in meters multiplied by the subject's height in meters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- 100, Salvador, Estado de Bahia, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from one study center in Brazil.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- TIV (18 to ≤ 60 Years): Healthy adult subjects 18 to ≤ 60 years who received one dose of trivalent, surface antigen inactivated subunit influenza virus vaccine (TIV) formulation 2015 Southern Hemisphere.
- TIV (≥ 61 Years): Healthy adult subjects ≥ 61 years who received one dose of trivalent, surface antigen inactivated subunit influenza virus vaccine (TIV) formulation 2015 Southern Hemisphere.
Period: Overall Study
Arm/Group | TIV (18 to ≤ 60 Years) | TIV (≥ 61 Years)
Started | 63 | 63
Completed | 63 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TIV (18 to ≤ 60 Years) | TIV (≥ 61 Years) | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (11.0) | 69.3 (6.9) | 50.7 (20.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 52 | 107
  Male | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Single Radial Hemolysis (SRH) Areas ≥25mm^2, Against Each of Three Vaccine Strains After Receiving One Dose of TIV.
Description: Immunogenicity was assessed in terms of percentages of subjects in both age groups with SRH areas ≥25mm^2 against each of the three vaccine strains, three weeks after receiving one dose of TIV.
  The related European Committee for Medicinal Products for Human Use (CHMP) criterion for the assessment of immunogenicity is met if the percentage of subjects achieving post vaccination SRH areas ≥ 25mm^2 is >70% for adults aged 18 to ≤60 years and >60% for subjects aged ≥61 years.
Time Frame: Day 1 and Day 22 post vaccination
Population: The analysis was performed on the per-protocol population (PP).
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TIV (18 to ≤ 60 Years) | TIV (≥ 61 Years)
Number analyzed (Participants) | 63 | 62
Percentages of subjects
  A/H1N1 (Day 1) | 62 [49 to 74] | 52 [39 to 65]
  A/H3N2 (Day 1) | 51 [38 to 64] | 40 [28 to 54]
  B strains (Day 1) | 71 [59 to 82] | 61 [48 to 73]
  A/H1N1 (Day 22) | 98 [91 to 100] | 63 [50 to 75]
  A/H3N2 (Day 22) | 84 [73 to 92] | 73 [60 to 83]
  B strains (Day 22) | 94 [85 to 98] | 84 [72 to 92]

2. Primary Outcome: Percentages of Subjects With Seroconversion or Significant Increase in SRH Area, Against Each of Three Vaccine Strains After Receiving One Dose of TIV.
Description: Immunogenicity was assessed in terms of percentages of subjects in both age groups achieving seroconversion or significant increase by SRH area against each of the three vaccine strains, three weeks after receiving one dose of TIV.
  Seroconversion is defined as percentage of subjects with a pre vaccination SRH area ≤ 4mm^2 achieving a post vaccination SRH area ≥ 25mm^2. Significant increase is defined as percentage of subjects with a pre-vaccination SRH area > 4mm^2 achieving at least 50% increase in post vaccination SRH area.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if >40% for adults aged 18 to ≤60 years and >30% for subjects aged ≥61 years achieve seroconversion or significant increase in post-vaccination SRH areas.
Time Frame: Day 22 post vaccination
Population: The analysis was performed on the PP dataset
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TIV (18 to ≤ 60 Years) | TIV (≥ 61 Years)
Number analyzed (Participants) | 63 | 62
Percentages of subjects
  A/H1N1 | 46 [33 to 59] | 39 [27 to 52]
  A/H3N2 | 49 [36 to 62] | 47 [34 to 60]
  B strains | 48 [35 to 61] | 32 [21 to 45]

3. Primary Outcome: Geometric Mean Ratio (GMR) of Post Vaccination Versus Pre Vaccination Geometric Mean Area (GMAs), After One Dose of TIV.
Description: The antibody responses were evaluated in terms of GMRs of post vaccination GMAs to pre vaccination GMAs against each of the three vaccine strains, three weeks after receiving one dose of TIV.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if the GMR day 22/day 1 is >2.5 for adults aged 18 to ≤60 years and > 2.0 in for subjects aged ≥61 years.
Time Frame: Day 22/ Day1 post vaccination
Population: The analysis was performed on the PP dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | TIV (18 to ≤ 60 Years) | TIV (≥ 61 Years)
Number analyzed (Participants) | 63 | 62
Ratio
  A/H1N1 | 2.3 [1.79 to 2.95] | 1.58 [1.39 to 1.81]
  A/H3N2 | 2.48 [1.8 to 3.42] | 2.18 [1.59 to 2.99]
  B strains | 2.28 [1.75 to 2.98] | 1.72 [1.35 to 2.17]

4. Primary Outcome: Percentages of Subjects With Haemagglutination Inhibition (HI) Titers ≥40, Against Each of Three Vaccine Strains After Receiving One Dose of TIV.
Description: Immunogenicity was assessed in terms of percentages of subjects in both age groups with HI titers ≥40, against each of the three vaccine strains, three weeks after receiving one dose of TIV.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if the percentage of subjects achieving HI titers ≥ 40 is >70% for adults aged 18 to ≤60 years and >60% for subjects aged ≥61 years.
Time Frame: Day 1 and Day 22 post vaccination
Population: The analysis was performed on the PP dataset.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | TIV (18 to ≤ 60 Years) | TIV (≥ 61 Years)
Number analyzed (Participants) | 63 | 62
Percentages of Subjects
  A/H1N1 (Day 1) | 89 [78 to 95] | 90 [80 to 96]
  A/H3N2 (Day 1) | 79 [67 to 89] | 87 [76 to 94]
  B strains (Day 1) | 46 [33 to 59] | 40 [28 to 54]
  A/H1N1 (Day 22) | 100 [94 to 100] | 98 [91 to 100]
  A/H3N2 (Day 22) | 100 [94 to 100] | 100 [94 to 100]
  B strains (Day 22) | 92 [82 to 97] | 60 [46 to 72]

5. Primary Outcome: Percentages of Subjects With Seroconversion or Significant Increase in HI Antibody Titers After Receiving One Dose of TIV.
Description: Immunogenicity was assessed in terms of percentages of subjects in both age groups achieving seroconversion or significant increase in HI antibody titers after receiving one dose of TIV.
  Seroconversion is defined as percentage of subjects with a pre vaccination HI titer <10 and a post vaccination titer ≥40. Significant increase is defined as percentage of subjects with a pre vaccination HI titer ≥10 and at least a 4-fold increase in post vaccination HI antibody titers.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if >40% for adults aged 18 to ≤60 years and >30% for subjects aged ≥61 years achieve seroconversion or significant increase in post-vaccination HI titers.
Time Frame: Day 22 post vaccination
Population: The analysis was performed on the PP dataset.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | TIV (18 to ≤ 60 Years) | TIV (≥ 61 Years)
Number analyzed (Participants) | 63 | 62
Percentages of Subjects
  A/H1N1 | 44 [32 to 58] | 23 [13 to 35]
  A/H3N2 | 56 [42 to 68] | 55 [42 to 68]
  B strains | 44 [32 to 58] | 13 [06 to 24]

6. Primary Outcome: GMR of Post Vaccination Versus Pre Vaccination HI Antibody Titers, After Receiving One Dose of TIV.
Description: The antibody responses following one vaccination of TIV were evaluated in terms of GMRs of post vaccination against pre vaccination geometric mean HI titers against each of the three vaccine strains, three weeks after receiving one dose of TIV.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if the GMR day 22/day 1 is >2.5 for adults aged 18 to ≤60 years and > 2.0 for subjects aged ≥61 years.
Time Frame: Day 22/Day 1 post vaccination
Population: The analysis was performed on the PP dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | TIV (18 to ≤ 60 Years) | TIV (≥ 61 Years)
Number analyzed (Participants) | 63 | 62
Ratio
  A/H1N1 | 3.96 [2.76 to 5.67] | 2.01 [1.68 to 2.4]
  A/H3N2 | 6.78 [4.57 to 10] | 5 [3.65 to 6.86]
  B strains | 3.57 [2.68 to 4.74] | 1.68 [1.39 to 2.03]

7. Primary Outcome: Number of Subjects Reporting Local and Systemic Solicited Adverse Events (AEs) After Receiving One Dose of TIV.
Description: The number of adult and elderly subjects reporting solicited local and systemic AEs and other solicited AEs after receiving one dose of TIV are reported.
Time Frame: Day 1 to Day 4 post vaccination (including 30 mins)
Population: Analysis was done on the solicited safety set population i.e. all subjects who have post vaccination solicited local and systemic adverse event data.
Measure: Number; unit: Number of Subjects
Arm/Group | TIV (18 to ≤ 60 Years) | TIV (≥ 61 Years)
Number analyzed (Participants) | 63 | 63
Number of Subjects
  Local AEs (Type I) | 16 | 19
  Injection-site induration (Type I) | 4 | 8
  Injection-site erythema (Type I) | 4 | 7
  Injection-site ecchymosis (Type I) | 1 | 1
  Injection-site pain | 14 | 9
  Systemic AEs (Type I) | 18 | 16
  Shivering/chills | 2 | 4
  Myalgia | 6 | 4
  Arthralgia | 3 | 5
  Headache | 12 | 8
  Fatigue | 6 | 4
  Malaise | 1 | 2
  Fever ≥38.0°C | 2 | 2
  Other- Treatment of pain and|or fever | 1 | 9
  Other- Prevention of pain and|or fever | 0 | 3

8. Primary Outcome: Number of Subjects Reporting Unsolicited AEs After Receiving One Dose of TIV.
Description: The number of subjects in both age groups reporting any unsolicited AEs between Day 1 to Day 4 after receiving one dose of TIV.
Time Frame: Day 1 to Day 4 post vaccination
Population: Analysis was done on the unsolicited safety set population i.e., all subjects who have post vaccination unsolicited adverse event data.
Measure: Number; unit: Number of Subjects
Arm/Group | TIV (18 to ≤ 60 Years) | TIV (≥ 61 Years)
Number analyzed (Participants) | 63 | 63
Number of Subjects
  Any AE | 6 | 10
  At least Possibly related AE | 5 | 6

9. Primary Outcome: Number of Subjects Reporting Unsolicited AEs After Receiving One Vaccination of TIV.
Description: The number of subjects in both age groups reporting any unsolicited AEs (between Day 1 to 4), serious adverse events (SAEs), medically attended AEs, AEs leading to premature withdrawal (Day 1 to Day 22), after receiving one vaccination of TIV is reported.
Time Frame: Day 1 to Day 22 post vaccination
Population: Analysis was done on the unsolicited safety set population i.e all subjects who have post vaccination unsolicited adverse event data
Measure: Number; unit: Number of Subjects
Arm/Group | TIV (18 to ≤ 60 Years) | TIV (≥ 61 Years)
Number analyzed (Participants) | 63 | 63
Number of Subjects
  Any AE | 13 | 19
  At least Possibly related AEs | 5 | 6
  Any SAE | 0 | 0
  At least Possibly related SAEs | 0 | 0
  Medically attended AEs | 3 | 4
  AEs leading to discontinuation | 0 | 0
  Death | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study, up to 22 days.
Description: All solicited AEs and unsolicited AEs were collected from Day1 to Day 4; all unsolicited SAEs, medically attended AEs, AEs leading to withdrawal from the study were collected from Day 1 to Day 22. Solicited AEs were collected systematically and the unsolicited AEs were collected non-systemically.
Arm/Group | TIV (18 to ≤ 60 Years) | TIV (≥ 61 Years) | Total
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63 | 0/126
Other Adverse Events (participants affected / at risk) | 27/63 | 33/63 | 60/126
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TIV (18 to ≤ 60 Years) (N=63) | TIV (≥ 61 Years) (N=63) | Total (N=126)
CHILLS (General disorders) | 2 | 4 | 6
FATIGUE (General disorders) | 6 | 4 | 10
INJECTION SITE ERYTHEMA (General disorders) | 4 | 7 | 11
INJECTION SITE INDURATION (General disorders) | 4 | 8 | 12
INJECTION SITE PAIN (General disorders) | 14 | 9 | 23
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 5 | 8
MYALGIA (Musculoskeletal and connective tissue disorders) | 7 | 6 | 13
HEADACHE (Nervous system disorders) | 14 | 12 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No